CLINICAL TRIAL: NCT00546702
Title: Multicenter, Open, Non-Randomised Phase III Clinical Study of Efficacy and Safety of Insulin Glulisine (HMR1964) Injected Subcutaneously in Patients With Type 1 Diabetes Mellitus Using Also Insulin Glargine During 26 Weeks of Therapy
Brief Title: Glulisine + Lantus in Type I Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_3505
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Insuline Glulisine

SUMMARY:
To evaluate the efficacy (in terms of change HbA1c from baseline to endpoint) and safety (in terms of adverse events, clinical chemistry, lipids, hematology) of insulin glulisine (HMR 1964) in subjects with type I diabetes mellitus To evaluate the change in HbA1c at week 26, blood/glucose parameters, hypoglycemia, insulin dose in subjects with type I diabetes mellitus receiving HMR 1964 and insulin glargine.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women (>18 years) with type I diabetes mellitus (onset of diabetes under the age of 40)
* An HbA1c range of >6.5 - <11%
* And on multiple injection regimen (more than 1 year of continuous insulin treatment)
* Body mass index <35.

Exclusion Criteria:

* Active proliferative diabetic retinopathy
* Diabetes other than type I diabetes mellitus
* Pancreatectomised subjects
* Subjects who have undergone pancreas and or islet cell transplantats, requiring treatment with not permited drugs during the study, previous treatment (in the period not less than 1 month before the beginning of the trial) with insulin glargine
* Hypersensitivity to insulin
* Major systemic diseases
* Impaired hepatic or renal function

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2004-09; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Change of HbA1c. | from baseline to endpoint.

SECONDARY OUTCOMES:
Change in HbA1c. | from baseline (week 1) to weeks 12 and 26
Blood glucose parameters, hypoglycaemic episodes and dosage of the mealtime and basal insulins. | from baseline to endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Efremenkova, Study Director — Sanofi
Locations (1):
- Sanofi-aventis, Moscow, Russia